CLINICAL TRIAL: NCT06117813
Title: Efficacy and Safety of the Nu.T for Improving Impaired Stereopsis Caused by Intermittent Exotropia : Multi Center, Randomized, Single-blind (Evaluator), Prospective Confirmatory Study
Brief Title: Visual Perceptual Learning Based Digital Therapeutics for Stereopsis in Intermittent Exotropia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nunaps Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NNS-IXTS-01
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nu.T (Experimental): Nu.T, 5 times a week for 8 weeks.
  Interventions: Device: Nu.T
- No-treatment Control (Other): No-treatment was administered during control period.
  Interventions: Other: No-Treatment Control

INTERVENTIONS:
Device: Nu.T — Participants receive visual perceptual training using the Nu.T software.
  Arms: Nu.T
Other: No-Treatment Control — No-treatment was administered during control period.
  Arms: No-treatment Control

SUMMARY:
This study evaluates the efficacy and safety of visual perceptual learning for improving stereopsis in intermittent exotropia. Half of participants will receive visual perceptual training using the Nu.T. The other half will not receive any training because there is no standard treatment for decreased stereopsis in intermittent exotropia.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent Exotropia patients aged 6 to 15
* Patients with decreased stereopsis above 50 arc seconds in Titmus Dot Test
* Able to use the Virtual Reality(VR) device
* Patient or legally authorized representative has signed the informed consent form

Exclusion Criteria:

* Incomitant strabismus patient with impaired eye movement
* Patients with amblyopia (Maximal corrective vision of one eye is less than 0.8 or maximal corrective vision both eyes more than two lines of difference)
* History of ophthalmic surgery
* Patient who has undergone or is currently undergoing cover treatment within one month for the purpose of treating strabismus or amblyopia
* Scheduled for ophthalmic surgery during the clinical trial participation period (8 weeks in the treatment group as of the registration date, Maximum 16 weeks in the control group as of the registration date)
* Difficult to understand and perform the stereopsis test.
* Abnormal Retinal Correspondence
* Patient with neurological abnormalities other than strabismus
* History of premature birth
* Participating in other clinical trial
* Any other condition that, in the opinion of the investigator, precludes participation in the trial

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Changes in (log) arc second of stereopsis from Baseline to 8 weeks | 8 weeks
  Stereopsis will be evaluated by a Titmus Dot Test.

SECONDARY OUTCOMES:
Proportion of subjects showing improved stereopsis at 8 weeks compared to baseline | 8 weeks
  Improved stereopsis means more than 2 steps increase in Titmus Dot Test.
Changes of Stereopsis based on Titmus Symbol Test from baseline to 8 weeks | 8 weeks
  Stereopsis will be evaluated by Titmus Symbol Test.
Changes of Stereopsis based on Distance Randot Stereotest from baseline to 8 weeks | 8 weeks
  Stereopsis will be evaluated by Distance Randot Stereotest.
Changes of strabismus angle from baseline to 8 weeks | 8 weeks
  Strabismus angle will be evaluated by distance and near-field.
Changes of convergence capability score from baseline to 8 weeks | 8 weeks
  Convergence capability will be evaluated in distance and near-field by LACTOSE System. The scores by LACTOSE System range from 0 to 4.
Changes of visuo-motor function from baseline to 8 weeks. | 8 weeks
  Visuo-motor function will be evaluated by the Bruininks-Oseretsky Test of Motor Proficiency Second Edition (BOT-2) test.

CONTACTS AND LOCATIONS:
Overall Officials: Yeji Moon, MD, PhD, Study Chair — Asan Medical Center
Locations (6):
- South Korea (6):
  - Inje University Ilsan Paik Hospital, Goyang
  - Hangil Eye Hospital, Incheon
  - Asan Medical Center, Seoul
  - Konkuk University Hospital, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Uijeongbu Eulji Medical Center, Eulji University, Uijeongbu-si